CLINICAL TRIAL: NCT03794141
Title: Effects of ApoE4 Genotype Information and Intervention Intensity on the Fulfillment of Lifestyle Changes and Sensory Preferences
Brief Title: Genetic Information as a Life Style Change Motivator
Acronym: APOE4MOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Natural Resources Institute Finland (Other Government)
Collaborators: University of Turku (Other); University of Eastern Finland (Other); Academy of Finland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 41007-00040400
Record Dates: First submitted 2018-12-13; First posted 2019-01-04 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2018-12

CONDITIONS: Health Behavior; Alzheimer Disease, Protection Against
MeSH Terms: conditions — Health Behavior; Alzheimer Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tervas (Experimental): Follow up group from an earlier study. Information on risk gene status. All test persons were given information on healthy diet and life style.
  Interventions: Behavioral: information on the risk gene status; Behavioral: life style advise
- Informed (Experimental): Information on risk gene status was given before intervention. All test persons were given information on healthy diet and life style.
  Interventions: Behavioral: information on the risk gene status; Behavioral: life style advise
- non informed (Active Comparator): Information on risk gene status was not given before intervention. All test persons were given information on healthy diet and life style.
  Interventions: Behavioral: life style advise

INTERVENTIONS:
Behavioral: information on the risk gene status — information on risk gene status (APOE4 allele or not) was given before intervention
  Arms: Informed; Tervas
Behavioral: life style advise — all test persons were given information on healthy diet and life style

SUMMARY:
The study investigates whether information on having a risk genotype (ApoE4) and life style advisory information affects lifestyle changes and sensory preferences. The project studies also the ethic aspects of giving the information of risk genotype.

DETAILED DESCRIPTION:
We will run intervention based on our earlier pilot study. It includes intensive intervention and a modification of our earlier pilot intervention. Our intervention methods are general lectures of the effects of healthy diet (Finnish Nutrition Recommendations 2014) and healthy lifestyle for all participants. Effects on motivation, attitudes and preferences will be studied and verified by questionnaires and risk factors of cardiovascular disease and Alzheimer disease by analyzing clinical markers of lipid metabolism, general phenotype markers and profiles of nutritional markers. Nutritional biomarkers will verify also the self-reported changes of diet in the questionnaires and in digital food diaries.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 60 years
* overall good health (no chronic conditions e.g. mental disorders, cancer, liver or kidney disease, current or previous diagnosis),
* body mass index (BMI) under 35 kg/m2,
* blood pressure under 140/90 mmHg (medication allowed),
* serum total cholesterol under 7.25 mmol/l (medication allowed)
* fasting plasma glucose level under 7 mmol/l.

Exclusion Criteria:

* Abnormal values of the alanine amino transferase, alkaline phosphatase, haptoglobin and thyroid stimulating hormone

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 333 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with good quality of dietary fat | 2 years
  A questionnaire according to Finnish guidelines of Suomen Sydänliitto ry, Helldán & Helakorpi, (2015)
Dietary habits, number of participants | 2 years
  A questionnaire asking for
  * Fish intake at least twice per week
  * Consumption of high fat and sugar foods
  * Consumption of vegetables
  * Alcohol consumption
  * Physical activity at least twice per week
Food choice questionnaire, health and taste attitude | 2 years
  Scale 1-7 (7 most important, fully agree)
Food involvement and Food mavenism, scale 1-5 | 2 years
  5 fully agree
Health concern, scale 1-9 | 2 years
  1 not concerned at all
Life-orientation test, scale 1-5 | 2 years
  1 fully agree
Locus of Control, state-trait anxiety inventory, Three-Factor Eating Questionnaire (TFEQ) scale 1-4 | 2 years
  4 fully agree
weight kg | 2 years
height m | 2 years
Waist circumference, cm | 2 years
Visceral fat level (1-30) | 2 years
blood pressure, mmHg | 2 years
Serum lipid levels mmol/L | 2 years
Blood glucose levels, mmol/L | 2 years
Serum lipid peroxidation, MDA/µM | 2 years
Serum Sensitive C reactive protein, mg/L | 2 years
Serum Hemoglobin, g/L | 2 years
Serum Alkaline phosphatase, U/L | 2 years
Serum Alanine aminotransferase, U/L | 2 years
Serum haptoglobin, g/L | 2 years
Plasma thyrotropin, mU/L | 2 years
serum APOE protein, mg/L | 2 years
serum brain-derived neurotrophic factor, ng/ml | 2 years
serum Fatty acids, g/100g fatty acids | 2 years
serum Carotenoids, retinol and α-tocopherol, Plasma total phenolics ng/µl | 2 years
Blood cell count | 2 years
APOE and BDNF genotype | baseline

SECONDARY OUTCOMES:
Body mass index | 2 years
  weight and height will be combined to report BMI in kg/m^2

CONTACTS AND LOCATIONS:
Overall Officials: Raija Tahvonen, Prof, Study Director — Natural Resources Institute Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leskinen HM, Tringham M, Karjalainen H, Iso-Touru TK, Hietaranta-Luoma HL, Marnila PJ, Pihlava JM, Hurme T, Kankaanpaa SJ, Puolijoki H, Akerman K, Tanner L, Sandell M, Vahakangas K, Hopia A, Tahvonen R, Rokka LS. APOE Genotype Disclosure and Lifestyle Advice in a Randomized Intervention Study with Finnish Participants. J Nutr. 2021 Jan 4;151(1):85-97. doi: 10.1093/jn/nxaa316. PMID 33188400